CLINICAL TRIAL: NCT05243537
Title: QTc Intervals in Former Preterm/Extreme Low Birth Weight Infants: a Pooled Study Proposal
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S66020
Record Dates: First submitted 2022-01-12; First posted 2022-02-17 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Qt Interval; Preterm Birth
Keywords: QTc; ELBW neonates; preterms; pharmacovigilance
MeSH Terms: conditions — Premature Birth | interventions — epicatechin gallate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QTc time interval in former preterm neonates, or term born healthy controls: former preterms and healthy term controls are defined as described in the cohort as previously published (Salaets et al, Pediatr Res 2021; Gervais et al, Pediatr Res 2020; Bassareo et al, J Matern Fetal Neonatal Med 2011). This includes both the perinatal characteristics as well as the characteristics collected at assessment (pediatric age or young adulthood) In all cases, an ECG was collected at rest, and these individual values (preterm or healthy term controls will be pooled.
  Interventions: Other: ECG (diagnostic)

INTERVENTIONS:
Other: ECG (diagnostic) — ECG collection (once, at rest), in both cases and controls

SUMMARY:
Pooling effort to collect previously reported data on QTc time in former preterm neonates, and compare these data to controls. At present and based on a recently conducted systematic search, there are conflicting data on the potential QT interval prolongation (all Bazett) in former extreme low birth weight (ELBW, <1000 g) infants or preterms.

Consequently, if investigators truly want to assess the presence or absence of either a difference or a prolongation of QTc intervals in this specific population, pooling of published data is likely the most effective approach (potential number of cases = 24 + 49 + 93 = 166; potential number of controls in the same studies = 24 + 53 + 87 = 164), preferably based on individual data.

Although the sample is to a large extent pragmatic (as available), the investigators hereby aim to target the 5 ms QTc prolongation applied by the authorities (FDA, EMA) in paired healthy adult volunteer studies as 'golden' standard as primary outcome variable [EMA guideline, FDA guidance].

DETAILED DESCRIPTION:
Preterm birth and gestational age at birth are associated with an increased risk for cardiovascular morbidity and mortality. In a large population-based cohort study with an incidence of preterm birth of 5.4 %, the adjusted hazard ratio of all-cause mortality in former preterms (23-33 weeks) was 1.44 in young adulthood (<50 years), most pronounced for cardiovascular mortality (1.89), diabetes (1.98) and chronic lung disease (2.28). Interestingly, the increased death risk was found across gestational age up to the ideal term age (39-41 weeks), but most prominent for the most immature group.

Besides better understanding of the underlying mechanisms associated with the 'Barker' and 'Brenner' cardiovascular risk hypotheses, there is an obvious need to further explore biomarkers to detect potential higher risk besides the gestational age or birth weight to translate this knowledge to clinical practice or secondary prevention strategies.

In a recent meta-analysis on changes in the preterm heart from birth to young adulthood, it was concluded that former preterms have morphological and functional cardiac impairments, proportionally to the degree of prematurity. In contrast to the echocardiographic differences in left and right ventricular systolic functions in former preterm when compared to term controls, observations on electrocardiographic (ECG) findings are less conclusive. Whether preterm birth is associated with conduction or repolarization abnormalities later in life is less well explored.

At present and based on a recently conducted systematic search, there are conflicting data on the potential QT interval prolongation (all Bazett) in former extreme low birth weight (ELBW, <1000 g) infants (data reported chronological).

Bassareo et al. reported that corrected QT (QTc) intervals and QT dispersion (QTd) were significantly prolonged in 24 former ELBW cases compared to 24 term controls (mean, ± SD: 417, 23.6 versus 369, 19.5 ms, and 30.4, 14.1 versus 24.6, 8.2 ms, respectively) (age at assessment = 23.2, SD 3.3 years).

Gervais et al. could subsequently not confirm these findings in 49 preterm cases (<30 weeks) when compared to 53 term born controls. At rest, mean QTc were 408, ± 34 and 409, ±SD 31 ms respectively (age at assessment = 18-33 years). Post-hoc power calculations showed that this study had 80% power to detect a difference of at least 18 ms in QTc between the two groups.

Finally, based on the PREMATCH study (ClinicalTrials.gov NCT02147457, S 56577), data on QTc observations are also available. QTc and QTd were similar between 93 ELBW cases and 87 controls [409 (range 360-465) versus 409 (337-460); 40 (0-100) versus 39 (0-110)] ms. When expressed by mean and SD, 409 (23) ms in the full dataset, 409 (SD 22) in former ELBW cases, 409 (SD 24) in controls [Salaets et al, Pediatr Res 2022]. Age, height, weight or body mass index were not associated with the QTc interval, while female sex (median difference 11.4 ms) and lower potassium (r=-0.26) were associated with longer QTc interval. We could not observe any significant association between QTc interval and perinatal characteristics (age at assessment 8-14 years). Post hoc analysis showed that our study had a power of 90 % to detect a difference of 11,45 ms between both groups.

Consequently, if researchers truly want to assess the presence or absence of either a difference or a prolongation of QTc intervals in this specific population, pooling of published data is likely the most effective approach (potential number of cases = 24 + 49 + 93 = 166; potential number of controls in the same studies = 24 + 53 + 87 = 164), preferably based on individual data. Although the sample is to a large extent pragmatic (as available), the investigators hereby aim to target the 5 ms QTc prolongation applied by the authorities (FDA, EMA) in paired healthy adult volunteer studies as 'golden' standard as primary outcome variable [EMA guideline, FDA guidance]. In all 3 cohorts, perinatal characteristics (like gestational age, weight, or pre- or postnatal steroids) were explored on their potential impact on the QTc interval, but all cohorts were underpowered to draw firm conclusions, so that these analyses will be included as secondary analyses.

Descriptive statistics will be used to report on the pooled dataset, and will be reported by mean and standard deviation, or median and range, pending normal distribution characteristics or incidence (%), (cases and controls, or cases only, respectively).

Statistical analysis will be used (two-tailed or one-tailed) to explore the relation of the data to the underlying population(s), like Rank correlation, Mann Whitney U or t-test (cases to controls, and within cases respectively). Based on the individual cohorts published, it is reasonable to anticipate normal distribution.

Power exploration using Mann-Whitney-U tests at alfa = 0,05 In order to find a significant two-tailed difference of 5ms, with a power of 90 % and extrapolating from the data distribution of the Leuven cohort, it was estimated that 467 subjects are required in both case and control groups. Decreasing the power to 80 % still requires 349 subjects in each group. In order to find a significant one-tailed difference of 5ms, with a power of 90 % and using the data distribution of the Leuven cohort, it was estimated that 381 subjects are required in both case and control groups.

Decreasing the power to 80 % still requires 275 subjects in each group (when using the FDA and EMA criteria to exclude an increase of 5 ms in former preterm cases).

In order to find a significant two-tailed difference of 10ms, with a power of 90 % and extrapolating from the data distribution of the Leuven cohort, it was estimate 118 subjects are required in both case and control groups. Decreasing the power to 80 % requires 88 subjects in each group.

In order to find a significant one-tailed difference of 10ms, with a power of 90 % and using the data distribution of the Leuven cohort, it was estimated that 96 subjects are required in both case and control groups. Decreasing the power to 80 % requires 70 subjects in each group. Inversely, having 166 and 164 subjects in each group and extrapolating the Leuven distribution data, this will have 90 % power to significantly discriminate a difference of 8.43ms (two-tailed) or 7.60ms (one-tailed), or 80 % power to significantly discriminate a difference of 7.28ms (two-tailed) or 6.46ms (one-tailed). Due to differences in data distribution between the cohorts: the actual discriminative power will probably be lower (the Leuven cohort -used for this estimation- has the narrowest standard deviation, and the Italian cohort has a different mean).

The investigators intend to conduct a post hoc power analysis with a difference (hypothesis: the mean QTc is not >5 ms higher in former preterm neonates compared to controls).

ELIGIBILITY:
Inclusion Criteria:

* included as 'case' in one of the cohorts retrieved by a systematic search on QTc values in former preterm neonates compared to healthy controls, or.
* included a 'control' in one of the cohorts retrieved by a systematic search on QTc values in former preterm neonates compared to healthy controls.

Exclusion Criteria:

* not included as 'case' in any of the cohorts retrieved by systematic search on QTc values in former preterm neonates compared to healthy controls
* not included as 'control' in any of the cohorts retrieved by systematic search on QTc values in former preterm neonates compared to healthy controls

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — QTc interval is known to be different between both genders
Study Population: The Bassareo cohort, Gervais cohort and Salaets cohort have been described in the original papers. we intent to pool the individual data of these cohorts (all these cohorts were constructed based on probability sampling)
  Bassareo, P. P. et al. Significant QT interval prolongation and long QT in young adult ex-preterm newborns with extremely low birth weight. J. Matern. Fetal Neonatal Med. 24, 1115-1118 (2011).
  Gervais, A. S. et al. Electrocardiographic features at rest and during exercise in young adults born preterm below 30 weeks of gestation. Pediatr. Res. 88, 305-311 (2020).
  Salaets, T. QTc intervals are not prolonged in former ELBW infants at pre-adolescent age. Pediatr. Res. 2021, online.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
QTc time interval | 1 year
  QTc time interval (in msec) in former preterms or healthy term controls

CONTACTS AND LOCATIONS:
Overall Officials: karel allegaert, MD, PhD, Principal Investigator — UZ Leuven
Locations (2):
- University Hospitals Leuven, Leuven, Belgium
- Centre Hospitalier Universitair Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
as part of the agreement, the individual data remain the ownership of the individual contributing centers, so that both centers should be contacted. This will be facilitated by the coordinating investigator (karel allegaert, karel.allegaert@uzleuven.be) upon request.

REFERENCES:
- [Background] Gervais AS, Flahault A, Chan T, Bastien-Tardif C, Al-Simaani A, Cloutier A, Luu TM, Abadir S, Nuyt AM. Electrocardiographic features at rest and during exercise in young adults born preterm below 30 weeks of gestation. Pediatr Res. 2020 Aug;88(2):305-311. doi: 10.1038/s41390-020-0814-9. Epub 2020 Mar 2. PMID 32120379
- [Background] Bassareo PP, Fanos V, Puddu M, Cadeddu C, Balzarini M, Mercuro G. Significant QT interval prolongation and long QT in young adult ex-preterm newborns with extremely low birth weight. J Matern Fetal Neonatal Med. 2011 Sep;24(9):1115-8. doi: 10.3109/14767058.2010.543600. Epub 2011 Jan 10. PMID 21219107
- [Result] Salaets T, Raaijmakers A, Zhang ZY, Yu YL, Wei DM, Staessen JA, Allegaert K. QTc intervals are not prolonged in former ELBW infants at pre-adolescent age. Pediatr Res. 2022 Sep;92(3):848-852. doi: 10.1038/s41390-021-01877-w. Epub 2021 Dec 2. PMID 34857877
- [Derived] Vanthienen J, Petrov MV, Luu TM, Cloutier A, Raaijmakers A, Staessen JA, Zhang Z, Salaets T, Laenen A, Smits A, Nuyt AM, Flahault A, Allegaert K. The QTc-Bazett Interval in Former Very Preterm Infants in Adolescence and Young Adulthood is Not Different from Term-Born Controls. Drug Saf. 2023 Sep;46(9):897-904. doi: 10.1007/s40264-023-01335-y. Epub 2023 Jul 28. PMID 37505401